CLINICAL TRIAL: NCT06373887
Title: The Efficacy of Weight-loss Diet Decision-making Based on Initial Gut Metabolic Modules (GMMs)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2023-09-005A
Record Dates: First submitted 2024-04-16; First posted 2024-04-18 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Weight Loss
Keywords: Gut Microbiome; Weight Loss Diet
MeSH Terms: conditions — Weight Loss

STUDY DESIGN:
Intervention Model Description: To compare the weight-loss efficacy of different carbohydrate degradation status under two different diet arm (low carbohydrate or low fat diet) to evaluate the benefits of initial gut microbiota profiling in precision weight loss dietary interventions.
Masking Description: Single-blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low carbohydrate diet (Experimental)
  Interventions: Dietary Supplement: plant-based Low carbohydrate diet
- Low fat diet arm (Active Comparator)
  Interventions: Dietary Supplement: plant-based Low low fat diet

INTERVENTIONS:
Dietary Supplement: plant-based Low carbohydrate diet — In the research, the high, medium, low carbohydrate degradation subjects were randomized to either plant-based Low carbohydrate diet or low fat diet to loss weight.
  Arms: Low carbohydrate diet
Dietary Supplement: plant-based Low low fat diet — In the research, the high, medium, low carbohydrate degradation subjects were randomized to either plant-based Low carbohydrate diet or low fat diet to loss weight.
  Arms: Low fat diet arm

SUMMARY:
In recent years, the technology to detect the gut microbiome's function has become increasingly developed. GMMs are tools (GitHub - raeslab/GMMs: A manually curated database of human gut metabolic modules.) for describing metabolic pathways for linking microbial metabolic function to species associated with a single metabolite, helping to analyze the transcriptional characteristics and metabolic functions of each bacterium, and studying their role of the food chain in the ecosystem. According to our previous research, the group with good weight loss response (more than 10% body weight loss in 8 weeks) after low-carb diet intervention has higher Shannon's diversity and carbohydrate degradation activity test by GMMs, implying the deficiency of availability of energy sources may cause more weight changes.

Based on the above research, we designed a low-carb diet (rich in monounsaturated fatty acids) and a low-fat diet (whole grains) with the same calories as a means of weight loss. The primary purpose of this study is to evaluate the pre-GMM test for determines the weight loss benefit of the intervention diet. Furthermore, we try to found the possible mechanism of whether metabolites of microbiota (e.g. SCFA) could affect the immune cell change which modulates adipose tissue .

DETAILED DESCRIPTION:
Many studies have shown that dysbiosis of gut microbiota is related to obesity and metabolic diseases4. Since there are many clinical guidelines for weight loss dietary recommendations that have been developed, successful long-term weight loss was still a challenge due to the personal variation of multi-omics markers at baseline and distinct diet-host-microbiome interaction1,2. A recent study2 related to successful long-term weight loss has found that the baseline microbiota composition and energy utilized patterns are related to the efficacy of long-term weight loss; The population with higher respiratory quotient (RQ) at baseline had significantly more weight loss when participating in a low-carb weight loss diet, suggesting that individuals with carbs as their main energy source had greater weight loss benefits when reducing carb sources. In our previous study, we also found that after the intervention of a low-carb diet (LCD), the groups with better weight loss results had higher diversity at the baseline, and the groups with better weight loss showed more active carbohydrate degradation using gut metabolic modules (GMMs) analysis. In contrast, one study5 showed an increased abundance of the genus (Dialister) encoding carbohydrate-active enzymes gene was associated with unsuccessful body weight loss when intervening with a weight-loss diet enriched with carbohydrates (Volumetric Diet). According to a recent study2 comparing a low-carb diet (LCD) and low-fat diet (LFD) for long-term weight loss, the LCD with a higher ratio of monounsaturated fatty acid (MUFA): saturated fatty acid (SFA) showed a better weight-loss response, while LFD with whole grain carbohydrate had better weight-loss response than refined grain carbohydrate. However, the weight loss efficacy between two diet arm within people with different carb degradation activities at the baseline was still unclear.

So far, there are no studies that use microbiota GMMs analysis before deciding which diet to intervene. Therefore, our study aims to investigate whether pre-examination and then intervention can bring benefits to weight loss efficacy.

Before the two dietary interventions, fecal microbiota analysis will be conducted to understand the metabolic activity of carbohydrates and then determine whether to enter the low-carbohydrate group or the low-fat group. The participants in this study will be divided into two groups: one group will have their gut microbiota measured before receiving dietary treatment, while the other group will be randomly assigned to one of the two dietary groups. Finally, the weight loss benefits and changes in gut microbiota and related biochemical data between the two groups will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Patients with BMI >=24 overweight and obesity without chronic disease or medication use.

Exclusion Criteria:

* a) Medication history of diabetes, hypertension, dyslipidemia, and cardiovascular diseases within two months.

  b) Bodyweight change within three months before the study. (+4kg). c) Participate in weight loss programs in the preceding 12 months. d) Use ABX, PPI, NSAID, laxatives, oral contraceptives, and antipsychotics within two months.

  e) Previous operations history for managing obesity (bariatric procedures and gastric bypass operation).

  f) Current smoking: at least 20 monthly cigarettes for over half a year. g) Alcohol consumption (> two glasses per day). h) Pregnancy, breastfeeding, chronic kidney dis-ease, autoimmune, viral chronic diseases (hepatitis C, B, HIV, etc.), and neoplastic diseases.

  i) Consumption of vegetarian or unusual diets. The Institutional Review Board approved all study protocols at TVGH.

Ages: 20 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-04-10 (Estimated); Primary Completion 2024-11-29 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Body weight loss/fat mass loss | 2 weeks to 2 months

SECONDARY OUTCOMES:
microbiota change | 2 months

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Veterans General Hospital, Taipei, Beitou District, Taiwan

IPD SHARING:
Plan to Share IPD: No